CLINICAL TRIAL: NCT07254286
Title: A Phase 1 Open-Label, Randomized, Crossover Food Effect and Formulation Assessment for Icovamenib Capsule in Healthy Volunteers
Brief Title: Food Effect Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVALENT-121
Record Dates: First submitted 2025-10-10; First posted 2025-11-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Food Effect

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, randomized, single dose, up to 7-way crossover study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Regimen A (Experimental): A - icovamenib capsule 100mg in fasted state
  Interventions: Drug: Icovamenib
- Regimen B (Experimental): B - icovamenib capsule 100mg in the fed state (0.5 h after initiation of low-fat breakfast)
  Interventions: Drug: Icovamenib
- Regimen C (Experimental): C - icovamenib capsule 100mg in the fed state (1 h after initiation of a low-fat breakfast)
  Interventions: Drug: Icovamenib
- Regimen D (Experimental): D - icovamenib capsule 100mg in the fed state (0.5 h after initiation of a high-fat breakfast)
  Interventions: Drug: Icovamenib
- Regimen E (Experimental): E - icovamenib capsule 100mg in the fed state (1 h after initiation of a high-fat breakfast)
  Interventions: Drug: Icovamenib
- Regimen F (Experimental): F - icovamenib HPMC capsule 100mg in the fed state (0.5 h after initiation of a high-fat breakfast)
  Interventions: Drug: Icovamenib HPMC
- Regimen G (Experimental): G - icovamenib HPMC capsule 100mg in the fed state (1h after initiation of a high-fat breakfast)
  Interventions: Drug: Icovamenib HPMC
- Regimen H (Experimental): H - icovamenib HPMC capsule 100mg in the fed state (0.5 h after initiation of a low-fat breakfast)
  Interventions: Drug: Icovamenib HPMC
- Regimen I (Experimental): I - icovamenib HPMC capsule 100mg in the fed state (1 h after initiation of a low-fat breakfast)
  Interventions: Drug: Icovamenib HPMC

INTERVENTIONS:
Drug: Icovamenib — Investigational Product
  Other Names: BMF-219
  Arms: Regimen A; Regimen B; Regimen C; Regimen D; Regimen E
Drug: Icovamenib HPMC — Investigational Product
  Other Names: BMF-219 HPMC
  Arms: Regimen F; Regimen G; Regimen H; Regimen I

SUMMARY:
A phase 1 open-label, randomized, crossover food effect and formulation assessment for icovamenib capsule in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase 1, open-label, randomized, single dose, up to 7-way crossover study. It is planned to enroll 60 healthy male and female subjects. Subjects will be randomized to receive one of 5 sequences, with N=12 per sequence. Subjects will be dosed in a single residency period. This study is designed to evaluate the effect of meal time and fat content of food on the PK and safety of the icovamenib capsule and the icovamenib hydroxypropyl methylcellulose (HPMC) capsule formulation.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent and Compliance

1. Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures.
2. Must be willing and able to comply with all study requirements. Baseline Characteristics
3. Healthy males or non-pregnant, non-lactating healthy females.
4. Body mass index (BMI) of 18.0 to 27.0 kg/m2 as measured at screening.
5. HbA1c ≤ 5.6%.
6. Fasting glucose ≤ 99 mg/dL.

Exclusion Criteria:

Medical/Surgical History and Mental Health

1. Mean QTcF interval greater than 440 msec on triplicate ECGs. Use of prescription or over-the-counter (OTC) medications known to significantly prolong the QT or QTcF interval.
2. History of hypertension or untreated hypertension (systolic blood pressure (BP) >140 mmHg and/or diastolic BP >90 mmHg).
3. Known self or family history (first-degree relative) of multiple endocrine neoplasia Type 1.
4. History of stomach or intestinal surgery or resection (except appendectomy, hernia and/or cholecystectomy).

   Diagnostic assessments.
5. Clinically significant abnormal clinical chemistry, hematology, coagulation or urinalysis as judged by the investigator.
6. History or evidence of hepatitis C virus (HCV), or hepatitis B virus (HBV) infection or human immunodeficiency virus (HIV) at screening.
7. Estimated creatinine clearance (CLcr) of <90 mL/min.
8. AST, ALT or bilirubin > ULN at screening.
9. Prior Study Participation.
10. Subjects who have received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose.
11. Prior and Concomitant Medication.
12. Subjects who are taking, or have taken, any prescribed or OTC drug or herbal remedies (other than HRT/hormonal contraception and up to 4 g per day acetaminophen) in the 14 days before first study medication administration.
13. Currently dieting (formal weight loss program) and/or are currently using or have used within 2 months of screening any drugs for weight management.
14. Received prior menin inhibitor treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Every other day for a max of 2 weeks
  Tmax
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Every other day for a max of 2 weeks
  Cmax
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Every other day for a max of 2 weeks
  AUC (0-last)
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Every other day for a max of 2 weeks
  AUC (0-inf)
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Every other day for a max of 2 weeks
  T1/2
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Every other day for a max of 2 weeks
  MRT (0-inf)
Evaluate food effect and PK profile of icovamenib capsule formulation in fed and fasted states | Time Frame: Every other day for a max of 2 weeks
  Tlag

SECONDARY OUTCOMES:
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  Tmax
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  Cmax
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  AUC (0-last)
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  AUC (0-inf)
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  T1/2
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  MRT(0-inf)
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  Tlag
Evaluate food effect and PK profile of icovamenib HPMC capsule formulation in fed states | Every other day for a max of 2 weeks
  Clast
Assess safety and tolerability of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  Incidence of adverse events (AEs)
Assess safety and tolerability in vital signs of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  Blood pressure (mmHg)
Assess safety and tolerability in vital signs of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  Heart rate (beats per minute)
Assess safety and tolerability in ECG of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  Heart rate (beats per minute)
Assess safety and tolerability in ECG of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  PR interval (ms)
Assess safety and tolerability in ECG of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  QRS interval (ms)
Assess safety and tolerability in ECG of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  QT interval (ms)
Assess safety and tolerability in ECG of icovamenib as capsule and HPMC capsule | Every other day for a max of 2 weeks
  QTcF interval (ms)
Number of participants with abnormal physical examination | Every other day for a max of 2 weeks
  General appearance
Number of participants with abnormal laboratory test findings | Every other day for a max of 2 weeks
  Clinical chemistry such as alanine aminotransferase (U/L), aspartate aminotransferase (U/L), alkaline phosphatase (U/L), total bilirubin (mg/dL)
Number of participants with abnormal laboratory test findings | Every other day for a max of 2 weeks
  Hematology such as red blood cell (x 10^6/uL), white blood cell (x 10^3/uL), and platelet count (x 10^3/uL)
Number of participants with abnormal laboratory test findings | Every other day for a max of 2 weeks
  Coagulation such as fibrinogen (mg/dL), prothrombin time (s), international normalized ratio (no units)
Number of participants with abnormal urine test findings | Every other day for a max of 2 weeks
  Urinalysis such as color (no units), appearance (no units), pH (pH)

CONTACTS AND LOCATIONS:
Overall Officials: Biomea Fusion Inc., Study Director — Biomea Fusion Inc.
Locations (1):
- Quotient Sciences - Miami, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No